CLINICAL TRIAL: NCT06322784
Title: Effects of Dietary Fiber (Oat Bran) Intervention on Inflammation, Intestinal Flora, Disease Activity and Quality of Life in Patients With Rheumatoid Arthritis
Brief Title: DF(Oat Bran) Intervention on Inflammation, Intestinal Flora, Disease Activity and Quality of Life in Patients With RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LiJingjing
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; dietary fiber; mechanism
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Experimental group=1,Control Group=2,
Who Masked: Investigator
Masking Description: Researchers set blinding to reduce implementation bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 12 week Mediterranean diet+dietary fiber intervention
  Interventions: Dietary Supplement: Oat bran (dietary fiber)
- Control group (No Intervention): 12 week Mediterranean diet

INTERVENTIONS:
Dietary Supplement: Oat bran (dietary fiber) — Dietary fiber, known as the "seventh type of nutrients," refers to carbohydrate polymers that have health benefits for the human body, mainly derived from plant cell walls such as grains, fruits, and vegetables.Mediterranean cuisine is a dietary pattern
  Other Names: The mediterranean Diet
  Arms: Experimental group

SUMMARY:
The goal of this clinical trial is to test in Rheumatoid arthritis. The main question it aims to answer are:

* To verify the effect of dietary fiber supplementation on reducing the level of inflammation;
* To verify the effect of dietary fiber supplementation on improving disease activity and quality of life in patients with rheumatoid arthritis .To verify the effect of dietary fiber supplementation on regulating the production of anti-inflammatory short-chain fatty acid in the gut of patients with rheumatoid arthritis.

The experimental group was supplemented with dietary fiber for 12 weeks, and the control group was fed with the Mediterranean diet. Before and after the intervention, 1 tube of 3ml blood and 1 soybean-sized stool were taken and a questionnaire was made

DETAILED DESCRIPTION:
Rheumatic arthritis (RA) is caused by chronic inflammation and joint injury caused by imbalance of pro-and anti-inflammatory mediators in the joints. Studies have shown that dietary fiber (DF) can be fermented by gut bacteria into anti-inflammatory short-chain fatty acid that may reduce joint inflammation, relieve symptoms and improve quality of life. The subjects were Randomized controlled trial to supplement DF12W individually, the intervention group to supplement DF12W, and the control group to supplement DF12W with routine diet, the differences of disease activity (DAS28 score) , inflammatory markers (TNF-a, IL-6, Mir-146a, Treg, ESR, CRP, etc.) and quality of life (SF-36) between the two groups were compared. The changes of intestinal flora were examined to verify the hypothesis. This study laid a good scientific foundation for dietary recommendation of RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR classification criteria, with a course of ≥ 2 years, and no changes in anti rheumatic drugs within 8 weeks prior to intervention;
* Age: 18-75 years old;
* DAS28-ESR ≥ 2.6 points, and fully controlled and treated with medication during screening visits;
* Sign an informed consent form and be able to complete the experiment according to the protocol.

Exclusion Criteria:

* Patients with mental illness, cognitive impairment, severe heart, lung, brain failure, serious complications, pregnancy, or life-threatening diseases;
* Patients with severe visual or auditory impairment and inability to understand research information;
* During the past 8 weeks of treatment with disease modifying anti rheumatic drugs (DMARDs), patients with food intolerance, allergies, and unwillingness to consume the intervention food in the study;
* In the past 10 years, there has been a history of tumors and eating disorders (such as neurogluttony, anorexia, binge eating, etc.);
* Participated in other intervention studies in the past three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Disease activity score | 12 weeks
  Questionnaire evaluation,Higher scores mean worse results
Quality of life score | 12 weeks
  Health Assessment Questionnaire,Higher scores mean worse results

SECONDARY OUTCOMES:
Compliance of oat bran | 12 weeks
  Use the follow-up record table to record the patients were followed up weekly on how many packets they ate . One pack a day, up to 7 packs a week, the greater the number, the better the compliance
Inflammatory indicators :TNF- α | 12 weeks
  Inflammatory factors were detected by ELISA ,In pg/ml.
Inflammatory indicators:IL-6 | 12 weeks
  Inflammatory factors were detected by ELISA ,In pg/ml.
Inflammatory indicators :IL-10 | 12 weeks
  Inflammatory factors were detected by ELISA ,In pg/ml.
Inflammatory indicators: ESR | 12 weeks
  Inflammatory factors were detected by Weiss method,In mm/h.
Inflammatory indicators :CRP | 12 weeks
  Inflammatory factors were detected by One-way immunodiffusion assay,In mg/L
gut flora | 12 weeks
  Metagenesis is used to detect intestinal flora, InTags Per Million
Adjustment of anti rheumatic drugs | Week 12
  The increment and decrement are unchanged.Incremental means going from not taking a synthetic anti-rheumatic drug to taking a synthetic anti-rheumatic drug, or increasing the dose of the original drug, or increasing the type of drug, or from the original traditional synthesis of disease-improving anti-rheumatic drugs adjusted for the biological synthesis of disease-improving anti-rheumatic drugs. A reduction in the dose of a synthetic anti-rheumatic drug is defined as a reduction in the dose of a synthetic anti-rheumatic drug from taking it to discontinuing it, or a reduction in the dose of the original drug, or from the original bio-synthesis to improve the condition of anti-rheumatic drugs adjusted to traditional synthesis to improve the condition of anti-rheumatic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Li, Master, Study Chair — Shenzhen People's Hospital
Locations (1):
- Jingjing Li, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Durholz K, Hofmann J, Iljazovic A, Hager J, Lucas S, Sarter K, Strowig T, Bang H, Rech J, Schett G, Zaiss MM. Dietary Short-Term Fiber Interventions in Arthritis Patients Increase Systemic SCFA Levels and Regulate Inflammation. Nutrients. 2020 Oct 20;12(10):3207. doi: 10.3390/nu12103207. PMID 33092271
- [Result] Yoshida Y, Tanaka T. Interleukin 6 and rheumatoid arthritis. Biomed Res Int. 2014;2014:698313. doi: 10.1155/2014/698313. Epub 2014 Jan 12. PMID 24524085
- [Result] Troeng T. [Medical decisions--theories for practical use?]. Lakartidningen. 1988 Sep 21;85(38):3081. No abstract available. Swedish. PMID 3199948
- [Result] Pauley KM, Satoh M, Chan AL, Bubb MR, Reeves WH, Chan EK. Upregulated miR-146a expression in peripheral blood mononuclear cells from rheumatoid arthritis patients. Arthritis Res Ther. 2008;10(4):R101. doi: 10.1186/ar2493. Epub 2008 Aug 29. PMID 18759964
- [Result] Bergot AS, Giri R, Thomas R. The microbiome and rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2019 Dec;33(6):101497. doi: 10.1016/j.berh.2020.101497. Epub 2020 Mar 19. PMID 32199713
- [Result] Horta-Baas G, Romero-Figueroa MDS, Montiel-Jarquin AJ, Pizano-Zarate ML, Garcia-Mena J, Ramirez-Duran N. Intestinal Dysbiosis and Rheumatoid Arthritis: A Link between Gut Microbiota and the Pathogenesis of Rheumatoid Arthritis. J Immunol Res. 2017;2017:4835189. doi: 10.1155/2017/4835189. Epub 2017 Aug 30. PMID 28948174
- [Result] Liu X, Zou Q, Zeng B, Fang Y, Wei H. Analysis of fecal Lactobacillus community structure in patients with early rheumatoid arthritis. Curr Microbiol. 2013 Aug;67(2):170-6. doi: 10.1007/s00284-013-0338-1. Epub 2013 Mar 13. PMID 23483307
- [Result] Zhang X, Zhang D, Jia H, Feng Q, Wang D, Liang D, Wu X, Li J, Tang L, Li Y, Lan Z, Chen B, Li Y, Zhong H, Xie H, Jie Z, Chen W, Tang S, Xu X, Wang X, Cai X, Liu S, Xia Y, Li J, Qiao X, Al-Aama JY, Chen H, Wang L, Wu QJ, Zhang F, Zheng W, Li Y, Zhang M, Luo G, Xue W, Xiao L, Li J, Chen W, Xu X, Yin Y, Yang H, Wang J, Kristiansen K, Liu L, Li T, Huang Q, Li Y, Wang J. The oral and gut microbiomes are perturbed in rheumatoid arthritis and partly normalized after treatment. Nat Med. 2015 Aug;21(8):895-905. doi: 10.1038/nm.3914. Epub 2015 Jul 27. PMID 26214836
- [Result] Liu X, Zeng B, Zhang J, Li W, Mou F, Wang H, Zou Q, Zhong B, Wu L, Wei H, Fang Y. Role of the Gut Microbiome in Modulating Arthritis Progression in Mice. Sci Rep. 2016 Aug 2;6:30594. doi: 10.1038/srep30594. PMID 27481047
- [Result] Skoldstam L, Hagfors L, Johansson G. An experimental study of a Mediterranean diet intervention for patients with rheumatoid arthritis. Ann Rheum Dis. 2003 Mar;62(3):208-14. doi: 10.1136/ard.62.3.208. PMID 12594104
- [Result] Turesson Wadell A, Barebring L, Hulander E, Gjertsson I, Hagberg L, Lindqvist HM, Winkvist A. Effects on health-related quality of life in the randomized, controlled crossover trial ADIRA (Anti-inflammatory Diet In Rheumatoid Arthritis). PLoS One. 2021 Oct 14;16(10):e0258716. doi: 10.1371/journal.pone.0258716. eCollection 2021. PMID 34648598
- [Result] Davis C, Bryan J, Hodgson J, Murphy K. Definition of the Mediterranean Diet; a Literature Review. Nutrients. 2015 Nov 5;7(11):9139-53. doi: 10.3390/nu7115459. PMID 26556369